CLINICAL TRIAL: NCT02595541
Title: Effects of Adding Oral Sildenafil to Intravenous Milrinone on Postoperative Pulmonary Hypertension in Pediatric Undergoing Repair of Ventricular Septal Defect
Brief Title: Oral Sildenafil and Intravenous Milrinone on Postoperative Pulmonary Hypertension
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esam Eldin Mohamed Abdalla, lecturer-college of medicine, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB000087140
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Pulmonary Hypertension
Keywords: pediatric; cardiac; sildenfil; milrinone; pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Milrinone; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- milrinone group (Active Comparator): milrinone
  Interventions: Drug: milrinone
- sildenafil and milrinone group (Active Comparator): milrinone and sildenafil
  Interventions: Drug: milrinone; Drug: Sildenafil

INTERVENTIONS:
Drug: milrinone — IV milrinone (0.75 mcg/kg) loading dose over one hour started during re-warming of the patient (before weaning from CPB) and followed by a maintenance dose of 0.75 mcg/kg/minutes till the end of the study.
  Other Names: primacor
Drug: Sildenafil — IV milrinone (0.75 mcg/kg) loading dose over one hour started during re-warming of the patient (before weaning from CPB) and followed by a maintenance dose of 0.75 mcg/kg/minutes till the end of the study. After baseline measurements, sildenafil (1mg/kg) administered in ICU via a nasogastric tube, to be repeated every 4 hours via a nasogastric tube or orally. Sildnafil is presented in tablet form which was dissolved in water to make a concentration of 1 mg/ml.
  Other Names: viagra
  Arms: sildenafil and milrinone group

SUMMARY:
Pulmonary hypertension (PH) is a consequence of an increase in pulmonary vascular resistance (PVR), pulmonary blood flow, pulmonary venous pressure, or a combination of these elements. Pulmonary arterial hypertension is a frequent complication of congenital heart disease, particularly in patients with systemic-to-pulmonary shunts. Persistent exposure o f the pulmonary vasculature to increased blood flow and pressure may result in vascular remodeling and dysfunction. This leads to increased pulmonary vascular resistance and, ultimately, to reversal of the shunt and development of Eisenmenger's syndrome. It may be more appropriate to define pulmonary hypertension according to the ratio of MPAP to mean systemic arterial pressure (MPAP/MAP) because children may have a low mean systemic blood pressure. MPAP/MAP ratio of < 0.25 is normal, a ratio of 0.33-0.5 indicates moderate pulmonary hypertension, and a ratio of > 0.5 is indicative of severe pulmonary hypertension

DETAILED DESCRIPTION:
30 Patients were randomly allocated in two equal groups; group MS (received intravenous milrinone and oral sildenafil) and group M (received only intravenous milrinone). Demographic data, patient's clinical data and different intraoperative times were recorded. In 1st postoperative 24 hours, we recorded; hemodynamic parameters [mean pulmonary arterial pressure (MPAP), mean systemic arterial pressure (MAP), heart rate, central venous pressure]. We calculated MPAP/MAP and inotropic score. The incidence of pulmonary hypertensive crisis, side effects of studied drugs and complications related to pulmonary artery catheter were recorded.

ELIGIBILITY:
Inclusion Criteria:

- Thirty patients in the age range 2-24 months scheduled for surgical closure of ventricular septal defect (VSD) associated with postoperative pulmonary hypertension [diagnosed in all patients by preoperative echocardiography and confirmed invasively by the pulmonary catheter before transfer to ICU by Mean Pulmonary Arterial Pressure (MPAP) > 25 mmHg or Mean Pulmonary Arterial Pressure (MPAP) /Mean Systemic Arterial Pressure (MAP) > 0.33] were enrolled in this study.

Exclusion Criteria:

* Patients with pre-existing obstructive lung disease, mitral valve disease, left ventricular dysfunction, and patients receiving preoperative pulmonary vasodilators

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
mean pulmonary arterial pressure | within the first 24 hours postoperative

SECONDARY OUTCOMES:
mean systemic blood pressure | within the first 24 hours postoperative
pulmonary hypertensive crisis | within the first 4 days postoperative